CLINICAL TRIAL: NCT01249976
Title: Evaluation of Recent Techniques for Diagnosing Central Venous Catheter-related Bloodstream Infections in Critically Ill Children
Brief Title: Recent Techniques for Diagnosing Central Venous Catheter-related Bloodstream Infections in Children
Acronym: Incat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K060210; N° ID RCB :2006-A000515-46 (Other: AFSSAPS)
Record Dates: First submitted 2010-11-27; First posted 2010-11-30 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Catheter-related Bloodstream Infection
Keywords: blood culture; central venous catheter; acridine orange leucocyte cytospin test; semi-quantitative skin culture
MeSH Terms: interventions — Blood Culture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- catheter-spearing diagnostic methods (Experimental): experimental
  Interventions: Other: blood culture

INTERVENTIONS:
Other: blood culture — blood culture

SUMMARY:
Removal of a central venous catheter (CVC) is often useful to prove its responsibility in a bloodstream infection. To avoid unnecessary removal of CVC, some catheter-spearing diagnostic methods have been recently developed. The aim of the study is to evaluate three catheter-spearing diagnostic methods in critically ill children: 1) the measurement of the differential time to positivity between a blood culture drawn from a peripherical vein and another one drawn through the CVC; 2) the exam of a blood sample drawn for the CVC and stained by acridine orange leucocyte cytospin test; 3) the semi-quantitative skin culture of the area around the insertion site of the CVC.

DETAILED DESCRIPTION:
Samples for the three techniques described above will be collected from the children admitted in Pediatric Intensive Care Unit with a CVC for more than 48 hours and with clinical or biological signs of systemic infection. Any investigation required to determine the origin of the infection will be performed, according to physician's judgement. If the CVC is removed or changed on a guide wire, a quantitative culture of the distal segment will be performed.

All the patients with a bloodstream infection and sampled according to the protocol will be included for statistical analysis. The physician and an independent medical expert will analyse if the bloodstream infection is CVC-related or not, according to the reference standard, by analysis of the clinical and bacteriological data, blinded towards the three studied techniques. The most optimal threshold will be determined and the sensibility, the specificity, the positive and negative predictable value of the three techniques will be calculated. Then sensibility of these three techniques will be compared.

ELIGIBILITY:
Inclusion Criteria:

* age between 0 and 18 years.
* Presence of a Central Venous Catheter for more than 48h (excepted umbilical catheter or peripherally inserted central catheters)
* Presence of at least one clinical or biological sign of systemic infection
* Parents are informed of the protocol and don't refuse the inclusion
* Prior inclusion in this study for the same bloodstream infection

Exclusion Criteria:

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
the differential time to positivity | maximum 24 hours
  To determine the sensibility, the specificity, the positive and negative predictible value of the measurement of the differential time to positivity between a blood culture drawn from a peripherical vein and another one drawn through the CVC, compared to the reference standard

SECONDARY OUTCOMES:
acridine orange leucocyte cytospin test. | maximun 24 hours
  To determine the sensibility, the specificity, the positive and negative predictible value of two others catheter -spearing diagnostic methods, compared to the reference standard :
  - the exam of a blood sample drawn for the CVC and stained by acridine orange leucocyte cytospin test.
semi-quantitative skin culture | maximum 24 hours
  To determine the sensibility, the specificity, the positive and negative predictible value of two others catheter -spearing diagnostic methods, compared to the reference standard :
  - the semi-quantitative skin culture of the area around the insertion site of the CVC.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Lesage, Md, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France